CLINICAL TRIAL: NCT04103229
Title: Investigation of Two Different Types of Solution and Volume for Inflating Foley Catheter Balloon in Indwelling Urinary Catheterization
Brief Title: Urinary Leakage in the Indwelling Urinary Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe AKBIYIK (Other)
Responsible Party: Sponsor-Investigator, Ayşe AKBIYIK, Doctor of Philosophy (PhD) Research Assistant, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EGE.0.20.05.00/OY/784/313
Record Dates: First submitted 2019-09-22; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Urine Leakage in the Indwelling Urinary Catheterization
Keywords: Urine Leakage; Indwelling urethral catheter; silicone catheter; Saline; Balloon; Distilled water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 10 ml sterile distilled water (Experimental): The indwelling urinary catheterization was inflated with 10 ml sterile distilled water (SDW) of the balloon.
  Interventions: Procedure: The use of different types and volumes of solutions to inflate the catheter balloon
- 15 ml sterile distilled water (Experimental): The indwelling urinary catheterization was inflated with 15 ml sterile distilled water (SDW) of the balloon.
  Interventions: Procedure: The use of different types and volumes of solutions to inflate the catheter balloon
- 10 ml 0.9% sodium chloride (NaCL) (Experimental): The indwelling urinary catheterization was inflated with 10 ml 0.9% sodium chloride (NaCL) of the balloon.
  Interventions: Procedure: The use of different types and volumes of solutions to inflate the catheter balloon
- 15 ml 0.9% sodium chloride (NaCL) (Experimental): The IUC was inflated with 15 ml 0.9% sodium chloride (NaCL) of the balloon.
  Interventions: Procedure: The use of different types and volumes of solutions to inflate the catheter balloon

INTERVENTIONS:
Procedure: The use of different types and volumes of solutions to inflate the catheter balloon — In catheterization procedure, catheter balloon was inflated according to the type and amount of fluid appropriate to the group to which the patient was assigned.

SUMMARY:
In the indwelling urinary catheterization (IUC), urinary leakage may develop around the catheter in the following days of catheterization. The volume and type of fluid used to inflate the catheter balloon has the potential to be a factor in the development of this problem.

In this study, the investigators aimed to investigate the effect of the type and amount of fluid used in inflating the silicone foley catheter balloon on the development of urinary leakage around the catheter. In addition to purpose, the following questions were answered to determine the optimal solution type and volume in inflating the balloon:

* What was the incidence of urinary leakage in IUC?
* Was there a relationship between catheterization time and urine leakage?
* Was there a relationship between the type of fluid used to inflate the foley catheter balloon and urine leakage?
* Was there a relationship between the amount of fluid used to inflate the foley catheter balloon and urine leakage?

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years,
* Patients with indication for IUC (presence of order),
* Patients eligible for the use of a 18 Fr silicone foley catheter,
* Patients who did not have a problem that could affect prostate hypertrophy and/or urinary system miction.

Exclusion Criteria:

* In the study, if urine leakage occurred within 12 hours after catheterization, it was assumed that the leakage was caused by the size of the catheter, and these patients/patients were excluded from the study.

Min Age: 18 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 64 male and 64 female patients were included in the study.
Enrollment: 128 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Development of urine leakage around the catheter | through study completion, about three years
  Patients were followed up every 12 hours for the presence of urine leakage around the catheter. The presence of urine leakage was monitored by macroscopic examination, wetting of the diaper, and pH meter strip wrapped around the catheter. In addition, urine samples of the urine leakage were collected, and urine pH and leakage pH were compared.
  Participation of the patients in the study groups was continued until one or more of the following criteria met:
  Urinary leakage around the catheter, Termination of catheterization, Transferring the patient to another unit, Development of Exitus.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse AKBIYIK, PhD, Principal Investigator — İzmir Katip Çelebi University

IPD SHARING:
Plan to Share IPD: No